CLINICAL TRIAL: NCT05081401
Title: Innovating(IN) Shorter(S), All- Oral, Precised(P), Individualized(I) Treatment Regimen(RE) for Rifampicin Resistant Tuberculosis(INSPIRE-TB)
Acronym: INSPIRE-TB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSPIRE-TB
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Multidrug Resistant Tuberculosis; Rifampicin Resistant Tuberculosis; Pre-XDR-TB
Keywords: multidrug resistant tuberculosis; shorter treatment; all-oral regimen; PZA sensitivity
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — A(2)C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- A-SOC (Active Comparator): The control arm for fluroquinolones susceptible participants is the current standard of care oral regimen for RR-TB recommended by Chinese national guidelines. The SOC regimen comprise one or two group A drugs(bedaquiline or linezolid, moxifloxacin or levofloxacin) and one group B drug(clofazimine or cycloserine) along with other companion drugs.
  Interventions: Combination Product: Bdq(Lzd)+Lfx(Mfx)+Cfz(Cs)+Pto+E+H+Z
- A1 (Experimental): The experimental A1 arm in fluroquinolones susceptible participants is a 9-month regimen consisted of bedaquiline, linezolid, fluroquinolones(moxifloxacin or levofloxacin), cycloserine, clofazimine.
  Interventions: Combination Product: A1
- A2a (Experimental): The experimental A2a arm in fluroquinolones susceptible participants is a 9-month regimen consisted of bedaquiline, linezolid, fluroquinolones(moxifloxacin or levofloxacin), cycloserine, pyrazinamide. The dosage of linezolid is 600mg daily for 9 months.
  Interventions: Combination Product: A2a
- A2b (Experimental): The experimental A2b arm in fluroquinolones susceptible participants is a 9-month regimen consisted of bedaquiline, linezolid, fluroquinolones(moxifloxacin or levofloxacin), cycloserine, pyrazinamide. The dosage of linezolid is 600mg daily for 2 months.
  Interventions: Combination Product: A2b
- A2c (Experimental): The experimental A2c arm in fluroquinolones susceptible participants is a 9-month regimen consisted of bedaquiline, linezolid, fluroquinolones(moxifloxacin or levofloxacin), cycloserine, pyrazinamide. The dosage of linezolid is 600mg daily for 2 months and then 300mg daily for 7 months.
  Interventions: Combination Product: A2c
- A3 (Experimental): The experimental A3 arm in fluroquinolones susceptible participants is a 9-month regimen consisted of bedaquiline, linezolid, fluroquinolones(moxifloxacin or levofloxacin), clofazimide, pyrazinamide.
  Interventions: Combination Product: A3
- A4 (Experimental): The experimental A4 arm in fluroquinolones susceptible participants is a 9-month regimen consisted of bedaquiline, fluroquinolones(moxifloxacin or levofloxacin), clofazimide, cycloserine, pyrazinamide.
  Interventions: Combination Product: A4
- A5 (Experimental): The experimental A4 arm in fluroquinolones susceptible participants is a 9-month regimen consisted of fluroquinolones(moxifloxacin or levofloxacin), linezolid, clofazimide, cycloserine, pyrazinamide.
  Interventions: Combination Product: A5
- B-SOC (Active Comparator): In fluroquinolones resistant participants, the comparator is a locally approved standard of care long regimen which is consistent with local guidelines for treatment of RR-TB in China and WHO recommendations. The control arm contain bedaquiline, cycloserine, clofazimine, and linezolid. Treatment duration is 20 months, with a 6-month intensive phase and a 14-month continuation phase.
  Interventions: Combination Product: B-SOC
- B1 (Experimental): In fluroquinolones resistant participants, the arm B1 is a 9-month treatment regimen with a combination of five drugs: bedaquiline, cycloserine, clofazimine, linezolid, pyrazinamide.
  Interventions: Combination Product: B1

INTERVENTIONS:
Combination Product: Bdq(Lzd)+Lfx(Mfx)+Cfz(Cs)+Pto+E+H+Z — A-SOC: 4Bdq(Lzd)+Lfx(Mfx)+Cfz(Cs)+Pto+E+H+Z/5Lfx(Mfx)+Cfz(Cs)+E+Z During the intensive phase: Bedaquiline(Linezolid);Levofloxacin(Moxifloxacin) All treatment is taken orally
  Arms: A-SOC
Combination Product: A1 — 9Bdq(6m)+Fq+Lzd+Cs+Cfz
  Arms: A1
Combination Product: A2a — 9Bdq(6m)+Fq+Lzd(600mg)+Cs+Z
  Arms: A2a
Combination Product: A2b — 9Bdq(6m)+Fq+Lzd(2m)+Cs+Z
  Arms: A2b
Combination Product: A2c — 9Bdq(6m)+Fq+Lzd(600mg-300mg)+Cs+Z
  Arms: A2c
Combination Product: A3 — 9Bdq(6m)+Fq+Lzd+Cfz+Z
  Arms: A3
Combination Product: A4 — 9Bdq(6m)+Fq+Cfz+Cs+Z
  Arms: A4
Combination Product: A5 — 9Fq+Lzd+Cfz+Cs+Z
  Arms: A5
Combination Product: B-SOC — 6Bdq+Lzd+Cs+Cfz/14Lzd+Cfz+Cs
  Arms: B-SOC
Combination Product: B1 — 9Bdq(6m)+Lzd+Cs+Cfz+Z
  Arms: B1

SUMMARY:
The INSPIRE-TB study is a pragmatic, multicentre, randomised, controlled, non-inferiority open-label trial to evaluate the efficacy and safety of seven 9-month oral regimens compared to a 9-month standard of care (SOC) regimen in RR-TB participants susceptible to fluoroquinolones, and a bedaquiline-containing 9-month oral regimen compared to a 20-month conventional regimen in RR-TB participants resistant to fluoroquinolones

DETAILED DESCRIPTION:
RR-TB patients susceptible to fluoroquinolones are identified with the Xpert MTB/XDR assay (Cepheid; Sunnyvale, CA, USA). Experimental arms are seven oral regimens with a five-drug combination of the following: bedaquiline, linezolid, a fluoroquinolone (moxifloxacin or levofloxacin), cycloserine, clofazimine, and pyrazinamide.To minimize potential toxicity, each regimen includes no more than two major QT-prolonging drugs (bedaquiline, clofazimine, and moxifloxacin). Treatment duration of the experimental regimens is 9 months. A 2-month extension of treatment is allowed with the presence of cavities at month 9 or in case of a positive culture at month 2. Baseline molecular drug susceptibility test (DST) of pyrazinamide will be performed using whole gene sequencing (WGS) technique. The result of molecular DST of pyrazinamide will be interpreted by technical staff at central laboratory of Huashan Hospital, Fudan University. Once a participant is proved resistant to pyrazinamide by WGS results at baseline, pyrazinamide will be discontinued with no need for extra drug replacement. The control regimen for RR-TB patients susceptible to fluoroquinolones is the current SOC oral regimen recommended by the national guidelines.

Pre-XDR TB patients are identified with the Xpert MTB/XDR assay. The experimental arm is a 9-month regimen consisting of bedaquiline, cycloserine, clofazimine, linezolid, and pyrazinamide. Treatment extension to 11 months is allowed with the presence of cavities at month 9 or in case of a positive culture at month 2. Pyrazinamide will be discontinued from the study regimen if baseline molecular DST results reveal pyrazinamide resistance. The comparator is a conventional longer regimen (20 months) consistent with the national guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 16-75 years with weight over 30kg, regardless of HIV status;
2. Pulmonary TB with rifampicin resistance diagnosed with either WHO-approved rapid molecular diagnostic test or phenotype drug susceptibility test (within 60 days prior to randomisation) ;
3. Signed informed consent form (ICF).

Exclusion Criteria:

1. Known allergies, hypersensitivity, or contraindication to any of the study drugs as described in additional material;
2. Participants combined with central nervous system TB, tuberculous osteomyelitis or arthritis, hematogenous disseminated pulmonary TB;
3. Patients known to be pregnant or breastfeeding at the time of enrollment;
4. Patients who have received second-line MDR-TB treatment for 14 days or more prior to enrollment;
5. Patients in critical condition and expected survival is estimated by physician to be less than 12 weeks.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
a favorable outcome at the end of study | at 21 months after randomization
  A favorable outcome is defined by the absence of previous unfavorable, and the last two culture results are negative. These two cultures must be taken from respiratory samples collected on separate visits at least 7 days apart. The latest culture sample should be collected between month 21 and 23.

SECONDARY OUTCOMES:
The median time to sputum culture conversion | at 21 months after randomization
  Time from treatment initiation to the first of two consecutive negative sputum culture conversion without an intervening positive culture.
The proportion of participants with grade 3 or higher AEs, SAEs | at 21 months after randomization
  To compare the proportion of patients who experience grade 3 or greater adverse events (AE graded according to the Common terminology criteria for adverse events, version 5.0), during treatment or follow-up in safety population.
All-cause mortality and treatment relevant mortality | at 21 months after randomization
  To compare the death rate and treatment relevant death rate during treatment or follow-up in safety population.
The proportion of participants with treatment relevant SAEs | at 21 months post-randomization
  To compare the proportion of patients treatment relevant SAEs, during treatment or follow-up in safety population.
The proportion of participants with grade 3 or higher QTc prolongation | at 21 months after randomization
  To compare the proportion of patients treatment relevant SAEs, during treatment or follow-up in safety population.
The proportion of participants experiencing permanent drug discontinuation or replacement due to QTc prolongation | at 21 months after randomization
  To compare the proportion of patients experiencing permanent drug discontinuation or replacement due to QTc prolongation, during treatment or follow-up in safety population.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PHD, Principal Investigator — Huashan Hospital
Locations (5):
- China (5):
  - Guiyang Public Health Treatment Center, Guiyang, Guizhou
  - People's Hospital of Qiandongnan, Kaili, Guizhou
  - The Third People's Hospital of Liupanshui, Liupanshui, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No